CLINICAL TRIAL: NCT00811408
Title: Modulating the Expression of Oncoproteins of Papillomavirus (HPV) to Increase Radiosensitivity: a Phase I Study of Antiviral Agent Cidofovir and Chemoradiotherapy Therapy in Cervical Cancers
Brief Title: Cidofovir in Treating Patients With Stage IB, Stage II, Stage III, or Stage IVA Cervical Cancer Who Are Receiving Chemotherapy and Radiation Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000626799; IGR-CSET-2007/1297; IGR-HPV-RX; INCA-RECF-0813; EUDRACT-2007-005505-21
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2009-07

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: human papilloma virus infection; cervical squamous cell carcinoma; cervical adenocarcinoma; stage IB cervical cancer; stage II cervical cancer; stage III cervical cancer; stage IVA cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Papillomavirus Infections | interventions — Carboplatin; Cidofovir; Brachytherapy; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cidofovir
Genetic: protein expression analysis
Other: laboratory biomarker analysis
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs such as cidofovir may make tumor cells more sensitive to radiation therapy. Giving cidofovir together with radiation therapy and chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of cidofovir in treating patients with stage IB, stage II, stage III, or stage IVA cervical cancer who are receiving chemotherapy together with radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of cidofovir when given as a radiosensitizer in patients with stage IB-IVA cervical cancer undergoing concurrent chemoradiotherapy.

Secondary

* Evaluate the influence of treatment on the expression of mRNA codons in HPV oncoproteins E6 and E7.
* Determine the rate of local control.

OUTLINE: This is a dose-escalation study of cidofovir.

Patients receive cidofovir IV weekly for 2 weeks prior to beginning radiotherapy and then once biweekly during radiotherapy. Patients undergo external pelvic radiotherapy for 5 weeks. Beginning ≤ 2 weeks later, patients undergo utero-vaginal brachytherapy. Some patients may also undergo a second course of external radiotherapy to the parametrium and/or lymph nodes ≤ 3 days after brachytherapy. Patients also receive concurrent carboplatin IV once weekly during external radiotherapy and brachytherapy.

Biological expression of HPV oncoproteins E6 and E7 is analyzed during treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of squamous cell carcinoma or adenocarcinoma of the cervix

  * Stage IB2 (> 4 cm), II, III, or IVA disease
* No lumbo-aortic metastasis
* Initial tumor must be HPV-positive

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy > 3 months
* ANC > 2,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Transaminases < 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase < 1.5 times ULN
* Bilirubin < 1.5 times ULN
* Creatinine < 1.5 times ULN
* Creatinine clearance ≥ 55 mL/min
* Proteinuria < 2 g/L
* Not pregnant
* Negative pregnancy test
* No renal disease
* No concurrent active infection
* No prior or concurrent psychiatric illness
* No history of cancer except for basal cell carcinoma
* No other active infection or serious illness that would prevent the patient from receiving study treatment
* No known psychological, familial, social, or geographic reason that would preclude clinical monitoring

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy or chemotherapy
* More than 30 days since prior experimental drugs

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of cidofovir

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deutsch, MD — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France